CLINICAL TRIAL: NCT05611125
Title: Nursing-Driven Primary Palliative Care for Urban-Dwelling African Americans With Chronic Lung Disease
Acronym: Hillman
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Rita & Alex Hillman Foundation (Unknown)
Responsible Party: Principal Investigator, Jeannette Kates, Co-Principal Investigator, Thomas Jefferson University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 083-51020-U32301; #22G.350 (Other: Jefferson Institutional Review Board)
Record Dates: First submitted 2022-09-27; First posted 2022-11-09 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Individuals in the intervention group will undergo a series of two telehealth video visits and a series of survey assessments at baseline, 3, and 6 months.
  Interventions: Other: Telehealth Integrated Primary Care (TIPC)
- Control (No Intervention): Individuals in the control group will continue with their usual standard of care and undergo a series of survey assessments at baseline, 3, and 6 months.

INTERVENTIONS:
Other: Telehealth Integrated Primary Care (TIPC) — The TIPC model of intervention incorporates video visits across research clinicians and patients' existing care clinicians for more synergized and accessible care provision for a given clinical indication. The first TIPC visit will center around the patient setting care goals for themselves and their caregiver with the help of a palliative care physician. The second TIPC visit will focus on assessing goal attainment and also close the care loop between their existing care team, a research-appointed palliative care team, and their involvement in our study.
  Other Names: TIPC
  Arms: Intervention

SUMMARY:
In prior work, this research team developed a telehealth primary care model (TIPC), designed in close partnership with patients and clinicians to address a widespread increase in telehealth use during the COVID-19 pandemic. Researchers will test the TIPC intervention to assess palliative care (PC) support for patients with chronic obstructive pulmonary disease (COPD) among a population of urban-dwelling, African American (AA) persons over the course of 15 months.

The aims of this study are to 1) evaluate patient, caregiver, and clinical team perspectives of feasibility and acceptability of the TIPC model with urban-dwelling AAs with advanced COPD, and 2) explore the impact of TIPC intervention on knowledge and completion of advanced care planning (ACP) and on hospice and healthcare utilization patterns in the target population, as well as on additional quality of life (QOL) endpoints, and compare these between individuals participating in the intervention group and control group.

DETAILED DESCRIPTION:
African Americans with chronic lung disease (CLD) experience higher-cost, lower-quality care (i.e. more untreated symptoms, poorer provider communication, care inconsistent with practices, lower hospice enrollment) compared to their white counterparts. Uptake of PC and ACP is also substantially lower amongst AAs and other underrepresented minorities (URMs) due to disparate access to information and mistrust in the healthcare system as generated by systemic, structural racism. Additionally, there are existing gaps in Jefferson's own PC program as revealed by our team's preliminary research into the program's level of cultural literacy. Interviews with black, indigenous people of color (BIPOC) enrolled with Jefferson PC revealed issues of clinician color blindness, an increased need for family engagement, and gaps in considering race and relationship to black pain in PC delivery.

This study will enroll 20 patients from Jefferson's Center City campuses. Half of the participants will be given the TIPC intervention, the other half will be assigned as controls who will receive their usual standard of care. All participants will be assessed over 6 months to assess changes in outcomes. Specifically amongst intervention patients, researchers will evaluate implementation outcomes (feasibility, acceptability, satisfaction, intervention uptake) of TIPC intervention at intervention start, post-visit 2, and 6 months after. Both intervention and control participants will be assessed for knowledge of ACP at 3 and 6 months, and health-related QOL, and caregiver burden at baseline, 3 months and 6 months.

Researchers will also measure clinical outcomes amongst both intervention and control patients (advance care planning and healthcare proxy designation, hospice use, avoidable healthcare utilization events) over 6 months.

Researchers will directly reach out to several departments including: Department of Medicine (Division of Pulmonary, Division of Hospital Medicine, and Division of Internal Medicine), Department of Family and Community Medicine, and Department of Emergency Medicine to identify patients (and, as applicable, their designated caregivers) for recruitment.

Once potential participants are identified, research team members will screen for eligibility criteria using EPIC. Recruitment will continue for all patients and caregivers until the anticipated enrollment goal for each group are reached (10 intervention, 10 controls).

Follow-up phone calls will be made to those who have not responded at approximately 3-7 day intervals.

Intervention subjects will partake in 2 telehealth visits as a part of the TIPC model. The first visit between patient, caregiver, and PC specialist will facilitate a patient-centered consultation guided by The Serious Illness Conversation Guide and involving patient completion of several PC assessments (i.e. Palliative Performance Scale,). The second visit between patient, caregiver, PC specialist and a pulmonology clinician/nurse will involve collaborative PC plan development and management and modeling of PC skills in an MDT framework.

This research team has trained staff to assess digital literacy and access barriers amongst all research participants. They will guide patients through accessing MyChart, creating an email (if needed), and perform test telehealth visits with patients prior to the scheduled clinical telehealth visits. If a patient is not able to connect at the time of their scheduled telehealth visit, a team member will call them via phone to again assist, as needed. This research team has ample experience with this, having created and deployed both the Telehealth Task Force (TTF) in the Sidney Kimmel Cancer Center (overseen by Dr. Worster) and the DOT (Digital Onboarding Taskforce) (overseen by Dr. Rising).

Evaluation of patient outcomes of the TIPC model will be ongoing across 6 months. Implementation outcomes will be measured amongst intervention patients. Feasibility, acceptability, and satisfaction collected via self-report will be collected at TIPC implementation and post-visit 2. Intervention uptake measured via chart review for references to the patient's PC plan in clinical encounters and PC plan-based referrals/adoptions will be analyzed over 6 months post-intervention.

Clinical outcomes will be measured for both subjects and controls. Advance care planning and healthcare proxy designation will be collected over 6 months via chart review, hospice use will be collected over 6 months via chart review for hospice enrollment and length of stay (LOS), and avoidable healthcare utilization events will be collected over 6 months via chart review for ED visits, urgent care (non-scheduled) visits, hospitalizations, and LOS with 'chief complaints' collected for each participant.

Additional follow-up outcomes of knowledge of ACP will be collected at 3 and 6 months and health-related QOL, and caregiver burden will be collected at baseline, 3 and 6 months for both subjects and controls via self-reporting.

ELIGIBILITY:
Inclusion Criteria:

* COPD Diagnosis
* Age 18 years or older

Exclusion Criteria:

* Traumatic Brain Injuries
* Incarceration
* Homelessness
* Developmental disorders
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Feasibility, Acceptability, Satisfaction regarding TIPC intervention as Assessed by Survey | 6 months
  Participants in the intervention group will report their experience with the TIPC model via survey questions. Participants will indicate whether or not they strongly disagree, disagree, have no opinion, agree, or strongly agree with a series of statements asking them about their experience with TIPC intervention.

SECONDARY OUTCOMES:
Change in Knowledge of Advanced Care Planning (ACP) | 3 months
  Participants will report the extent to which participating in video visits improved their knowledge regarding ACP. This will be assessed via a single-item statement that participants will say they either strongly disagree, disagree, have no opinion on, agree, or strongly agree with.
Change in Knowledge of Advanced Care Planning (ACP) | 6 months
  Participants will report the extent to which participating in video visits improved their knowledge regarding ACP. This will be assessed via a single-item statement that participants will say they either strongly disagree, disagree, have no opinion on, agree, or strongly agree with.
Change in Disease-Specific Quality of Life as Assessed by the CCQ | Baseline
  Participants report their disease-specific quality of life (QOL) by utilizing the Clinical COPD Questionnaire (CCQ). The CCQ measures COPD-specific QOL & asks a variety of symptom-related questions. A summary index score is derived by applying an appropriate value set to the responses for each question (never/not limited at all=0, hardly ever/very slightly limited=0.1, a few times/slightly limited=0.2, several times/moderately limited=0.3, many times/very limited=0.4, a great many times/extremely limited=0.5, almost all the time/totally limited or unable to do=0.6). Pts can score up to 6 points with a higher score being negatively associated with a lower QOL.
Change in Disease-Specific Quality of Life as Assessed by the CCQ | 3 months
  Participants report their disease-specific quality of life (QOL) by utilizing the Clinical COPD Questionnaire (CCQ). The CCQ measures COPD-specific QOL & asks a variety of symptom-related questions. A summary index score is derived by applying an appropriate value set to the responses for each question (never/not limited at all=0, hardly ever/very slightly limited=0.1, a few times/slightly limited=0.2, several times/moderately limited=0.3, many times/very limited=0.4, a great many times/extremely limited=0.5, almost all the time/totally limited or unable to do=0.6). Pts can score up to 6 points with a higher score being negatively associated with a lower QOL.
Change in Disease-Specific Quality of Life as Assessed by the CCQ | 6 months
  Participants report their disease-specific quality of life (QOL) by utilizing the Clinical COPD Questionnaire (CCQ). The CCQ measures COPD-specific QOL & asks a variety of symptom-related questions. A summary index score is derived by applying an appropriate value set to the responses for each question (never/not limited at all=0, hardly ever/very slightly limited=0.1, a few times/slightly limited=0.2, several times/moderately limited=0.3, many times/very limited=0.4, a great many times/extremely limited=0.5, almost all the time/totally limited or unable to do=0.6). Pts can score up to 6 points with a higher score being negatively associated with a lower QOL.
Change in General Quality of Life as Assessed by the FACIT-Pal | Baseline
  Participants report their quality of life (QOL) by utilizing the Functional Assessment of Chronic Illness Therapy - Palliative Care (FACIT-Pal). FACIT-Pal measures areas that include physical, social/family, emotional, & functional well-beings. A summary index score is derived by applying an appropriate value set to the responses for each question (not at all=0, a little bit=1, somewhat=2, quite a bit=3, very much=4). Pts can score up to 184 points with a higher score being associated with a higher QOL.
Change in General Quality of Life as Assessed by the FACIT-Pal | 3 months
  Participants report their quality of life (QOL) by utilizing the Functional Assessment of Chronic Illness Therapy - Palliative Care (FACIT-Pal). FACIT-Pal measures areas that include physical, social/family, emotional, & functional well-beings. A summary index score is derived by applying an appropriate value set to the responses for each question (not at all=0, a little bit=1, somewhat=2, quite a bit=3, very much=4). Pts can score up to 184 points with a higher score being associated with a higher QOL.
Change in General Quality of Life as Assessed by the FACIT-Pal | 6 months
  Participants report their quality of life (QOL) by utilizing the Functional Assessment of Chronic Illness Therapy - Palliative Care (FACIT-Pal). FACIT-Pal measures areas that include physical, social/family, emotional, & functional well-beings. A summary index score is derived by applying an appropriate value set to the responses for each question (not at all=0, a little bit=1, somewhat=2, quite a bit=3, very much=4). Pts can score up to 184 points with a higher score being associated with a higher QOL.
Change in Caregiver Burden | Baseline
  Participating caregivers will explore how taking care of their loved ones has impacted their daily lives via the Caregiver Strain Index (CSI). The CSI measures areas that include but are not limited to sleep hygiene, convenience of care, physical strain, family adjustments as a result of care, financial burden, and more. A summary index score is derived by applying an appropriate value set to the responses for each question (yes=1, no=0). Patients can score up to 12 points with a score of 7 or higher being associated with a higher level of caregiver burden experienced.
Change in Caregiver Burden | 3 months
  Participating caregivers will explore how taking care of their loved ones has impacted their daily lives via the Caregiver Strain Index (CSI). The CSI measures areas that include but are not limited to sleep hygiene, convenience of care, physical strain, family adjustments as a result of care, financial burden, and more. A summary index score is derived by applying an appropriate value set to the responses for each question (yes=1, no=0). Patients can score up to 12 points with a score of 7 or higher being associated with a higher level of caregiver burden experienced.
Change in Caregiver Burden | 6 months
  Participating caregivers will explore how taking care of their loved ones has impacted their daily lives via the Caregiver Strain Index (CSI). The CSI measures areas that include but are not limited to sleep hygiene, convenience of care, physical strain, family adjustments as a result of care, financial burden, and more. A summary index score is derived by applying an appropriate value set to the responses for each question (yes=1, no=0). Patients can score up to 12 points with a score of 7 or higher being associated with a higher level of caregiver burden experienced.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT05611125/ICF_000.pdf